CLINICAL TRIAL: NCT07003594
Title: Effect of Education Given With Jigsaw IV Learning Technique for Physical Assessment of Heart and Thorax on Knowledge and Skills of Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17162298600-228
Record Dates: First submitted 2025-02-20; First posted 2025-06-04 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Nursing Education Research; Nursing Education

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention Group:They train with the Jigsaw IV technique.
  Interventions: Other: Jigsaw IV technique
- Control Group (No Intervention): Control Group: They are educated in the traditional way.

INTERVENTIONS:
Other: Jigsaw IV technique — The Intervention Group receives training in cardiothoracic examination using the Jigsaw IV technique.
  Arms: Intervention Group

SUMMARY:
Title: The Effect of Jigsaw IV Learning Technique on Nursing Students' Knowledge and Skills in Heart and Thorax Assessment Objective: This study aims to evaluate the impact of education using the Jigsaw IV learning technique on the knowledge and skills of nursing students in performing physical assessments of the heart and thorax.

Methodology: A randomized controlled trial will be conducted with 70 second-year nursing students at Baskent University. Participants will be divided into an intervention group (n=35), receiving Jigsaw IV-based education, and a control group (n=35), receiving traditional education. Data collection, scheduled between 22.02.2025 and 22.05.2025, will include a Personal Information Form, Pretest/Posttest for Knowledge Assessment, Skill Assessment Form, and Jigsaw Opinion Scale. Knowledge levels will be analyzed using an independent samples t-test, skill levels using the Mann-Whitney U test, and students' perceptions of the Jigsaw IV method through frequency and percentage analysis.

Expected Outcome:The study will assess whether the Jigsaw IV method enhances students' knowledge and skills in heart and thorax assessment, contributing to the evaluation of its effectiveness in nursing education.

ELIGIBILITY:
Inclusion Criteria:

* Being a 2nd year nursing student.

Exclusion Criteria:

* not volunteering to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-06-25 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Knowledge level for heart and thoracic examination | Before the application starts and 2 weeks after training with jigsaw IV
skill performance level for heart and thoracic examination | 2 weeks after training with jigsaw IV
Jigsaw Opinion Scale (JOS) | immediately after the intervention
  Jigsaw Opinion Scale (JGÖ) developed by Şimşek (2007) was used to determine the students' opinions about the Jigsaw method. The 14 items of JGÖ are in the 5-point Likert type as "Very Effective", "Somewhat More Effective", "Equally Effective", "Less Effective" and "Much Less Effective" for comparing the jigsaw technique with the traditional learning method. The fifteenth item is open-ended and evaluates the students' positive and negative opinions about the technique. The internal consistency coefficient of JGÖ was determined as 0.70 in the original study. The total Cronbach alpha coefficient of the scale for the sample group of this study was found to be 0.76.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No